CLINICAL TRIAL: NCT02066675
Title: SAFETY AND ACTIVITY OF TRABECTEDIN AS FIRST LINE IN ADVANCED SOFT TISSUE SARCOMA (STS) PATIENTS UNFIT TO RECEIVE STANDARD CHEMOTHERAPY: A PROSPECTIVE PHASE II STUDY WITH CLINICAL AND MOLECULAR CORRELATES
Brief Title: Trabectedin First Line Therapy In Unfit Sarcoma Study
Acronym: TR1US
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG TR1US; 2013-001467-23 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Metastatic and Locally Advanced Soft Tissue Tumor Patients Unfit to Receive; Standard Chemotherapy
Keywords: Metastatic; Locally advanced; Soft tissue tumors
MeSH Terms: conditions — Neoplasm Metastasis; Soft Tissue Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trabectedin (Experimental): Trabectedin administered at the dose of 1.5 mg/mq-1.3 mg/mq a 24-hour continuous infusion via a central venous access, every 3 weeks
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — Each patients will receive intravenous trabectedin (1.5 mg/mq-1.3 mg/mq) over 24 hours every 3 weeks
  Other Names: Yondelis

SUMMARY:
Phase II, non-randomized, two-stage study according to Bryant & Day The study enroll patients with Metastatic and locally advanced soft tissue sarcoma unfit to receive standard chemotherapy (doxorubicin/epirubicin and/or ifosfamide)

DETAILED DESCRIPTION:
Soft tissue sarcomas are a group of rare and aggressive disease, comprising more than a hundred different histological subtypes and mainly originating from the embryonic mesoderm. Today, they represent less than 1% of all adult cancers, with an incidence of 3/100000/year and a median age at diagnosis of 65 years. Despite the progress done in the last decade, approximately 50% of STS patients still develop distant metastases within 3 years from the diagnosis and die from their disease. Doxorubicin (or epirubicin) and ifosfamide have been proved to be active in the treatment of STS and they are widely used, alone or in combination, as a first line therapy for locally advanced and metastatic patients. However, the response rate to the combination regimen in non-pretreated patients does not exceed 30-40%, and large randomized clinical trials failed to demonstrate any advantage in survival for the combination compared to single-agent treatment. Trabectedin (Yondelis®) is a marine-derived anticancer agent that has been approved in the European Union as a single agent for the treatment of STS patients after failure of standard chemotherapy (doxorubicin and/or ifosfamide) or for those unsuited to receive these agents. Even if the response rate in soft tissue sarcoma does not exceed 10%, trabectedin can provide a significant clinical benefit, by arresting disease progression in almost 50% of treated patients, with a progression-free survival rate of 20% at 6 months. Trabectedin was found to be particularly active in the treatment of myxoid liposarcoma and uterine leiomyosarcoma, for which better results have been obtained in terms of response rate and survival, suggesting an histotype driven activity. The toxicity profile of trabectedin given as second line therapy has been widely assessed in clinical studies and was largely manageable, with the majority of adverse events being grade 1 or 2 toxicities, generally reversible, dose or time dependent and noncumulative. The good tolerability profile observed in the trials seems to be confirmed also in everyday clinical practice. Conversely, few data are available at the moment about tolerability profile for those patients treated with trabectedin as first line because of medical conditions contraindicating the use of standard agents. The aim of this phase II study is to assess and describe trabectedin toxicity profile in this subset of negatively selected advanced inoperable STS patients.

ELIGIBILITY:
Inclusion criteria

* Adult patients (≥18 years), who, in the judgment of the clinician, is deemed not suitable to receive an anthracycline and/or ifosfamide based chemotherapy;
* Pathological diagnosis of soft tissue sarcoma
* Inoperable, locally advanced or metastatic tumor;
* Unsuited to receive doxorubicine and ifosfamide: ie stable arrhythmia, previous myocardial infarction; age≥80 years
* Eastern Cooperative Oncology Group Performance Status 0-2
* Glomerular filtration rate ≥30 mL per min
* Adequate hematologic function: Hemoglobin ≥9 g/dL; Absolute neutrophil count ≥1,500/μL, and Platelet count ≥100,000/microliter
* Creatinine phosphokinase < 2.5 Upper Normal Limit
* Adequate hepatic function: total bilirubin < Upper Normal Limit, total alkaline phosphatase < 2.5 Upper Normal Limit, or if > 2.5 Upper Normal Limit consider alkaline phosphatase liver fraction or gamma-glutamyltransferase or 5' nucleotidase must be < Transminase <2.5 x Upper Normal Limit, Albumin > 20 g/L.
* Patient´s written informed consent

Exclusion criteria

* Prior exposure to Trabectedin
* Performance status ≥2.
* Prior treatment with anthracyclines and or ifosfamide.
* History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission for 5 or more years and judged of negligible potential of relapse.
* Active viral hepatitis or chronic liver diseases, which in the judgement of the primary investigator represents a clinical contraindication to the therapy.
* Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within 6 months before enrolment, uncontrolled arterial hypertension or arrhythmias, left ventricular ejection fraction <40%
* Active major infection.
* Other serious concomitant illnesses
* Pregnant subjects or breast feeding, or planning to become pregnant within 6 months after the end of treatment All sexually active female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the 7 days prior to enrollment and must agree to use highly effective contraception during treatment and for 6 months after the end of treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival Rate | 3 Months
  The primary end point of this trial is the Progression Free Survival Rate at 3 months Non progression, is defined as Complete Response, Partial Response or Stable Disease according to Response Evaluation Criteria In Solid Tumours v.1.1 criteria.

SECONDARY OUTCOMES:
Tolerability and intolerable adverse reaction rate. | Day21
  Intolerable toxicity is defined as every Adverse Events leading to treatment discontinuation or dose-reduction; furthermore, any Adverse Events of at least grade 3 not resolved within 3 weeks of appropriate management should be regarded as an intolerable toxicity event. For haematological toxicity, given that the use of growth factors will be allowed, an intolerable toxicity is defined either as any grade 4 event, or a grade 3 event not resolved with adequate treatment.
Objective response rate | 5 years
  Proportion of patients whose best response is either partial response or complete response
Progression free survival | Average of 5 Months
  It's the length of time during and after the treatment of a disease, that a patient lives with the disease but it does not progress
Overall survival | 18 Months (average)
  it's the length of time after the treatment's end that the patient survives

CONTACTS AND LOCATIONS:
Overall Officials: Federica Grosso, MD, Principal Investigator — ASO SS Antonio e Biagio e C Arrigo Alessandria, Italy
Locations (16):
- Italy (16):
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola, FC
  - Ospedale Galliera, Genova, Genovs
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST, Genova, GE
  - Ospedale Villa Scassi, Genova, GE
  - Ospedale Misericordia e Dolce" Istituto Toscano Tumori, Azienda USL4, Prato, PO
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - Presidio Sanitario Gradenigo, Torino, TO
  - A.S.O. "SS Antonio e Biagio e Cesare Arrigo", Alessandria
  - Istituti Ortopedici Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - Ospedale SS. Trinità di Sora, Frosinone
  - IST, Genova
  - Policlinico Federico II Napoli, Napoli
  - Istituto Oncologico Veneto, Padua
  - Ospedale Giaccone, Palermo
  - Campus Biomedico, Roma

REFERENCES:
- [Background] Fayette J, Coquard IR, Alberti L, Boyle H, Meeus P, Decouvelaere AV, Thiesse P, Sunyach MP, Ranchere D, Blay JY. ET-743: a novel agent with activity in soft-tissue sarcomas. Curr Opin Oncol. 2006 Jul;18(4):347-53. doi: 10.1097/01.cco.0000228740.70379.3f. PMID 16721129